CLINICAL TRIAL: NCT04810364
Title: Systemic Inflammation and Progression of Atherosclerosis in HIV Patients Underwent Noninvasive and Invasive Multimodality Imaging
Brief Title: HIV Infection And Evolvement of Atherosclerotic Plaque
Acronym: HIVE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Central Clinical Hospital of the Russian Academy of Sciences (Other Government)
Collaborators: Moscow Regional Centre For HIV Care and Prevention (Unknown)
Responsible Party: Sponsor
Other Study IDs: HIVE
Record Dates: First submitted 2021-03-12; First posted 2021-03-23 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Coronary Artery Disease; Atherosclerosis, Coronary; Hiv; HIV Infections; Stable Chronic Angina
Keywords: Coronary Angiography; Echocardiography; Markers of Inflammation; Lipid Profile; Percutaneous transluminal coronary angioplasty; Percutaneous coronary intervention; Coronary Artery Diseases; Atherosclerosis; HIV; Plaque burden; SYNTAX score; Fractional flow reserve; Optical coherence tomography; Intravascular ultrasound; Intravascular imaging
MeSH Terms: conditions — Coronary Artery Disease; Acquired Immunodeficiency Syndrome; HIV Infections; Angina, Stable; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Blood samples to test the main hypothesis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All HIV-positive patients with chronic coronary syndrome: The Group includes all HIV-positive patients with stable chest pain. The progression of atherosclerosis will be quantitatively characterized by the parameters of the lesions (e.g. plaque burden, cap thickness, arterial remodeling, presence of erosions or rupture, malaposition of the stent, a vessel injury score, etc.). The imaging data will be handled with expert-level post-processing software.
  Interventions: Radiation: Quantitative coronary angiography, intravascular imaging with percutaneous intervention

INTERVENTIONS:
Radiation: Quantitative coronary angiography, intravascular imaging with percutaneous intervention — Coronaries will be shot with AXIOM Artis dFC (Siemens, Munich,Germany) or systems from any other vendors. In case if necessary the procedure will be delayed for intravascular imaging (OCT, IVUS, VH-IVUS, NIRS) and/ or percutaneous intervention (with implantation of the medical device).
  Other Names: QCA; Coronary intravascular imaging

SUMMARY:
In a prospective multi-center observational study, 200 HIV-infected patients treated with antiretroviral treatment (ART) and who suffered from coronary artery disease (CAD) will be enrolled. Blood samples for biological parameters will be collected with all participants: lipid profile and markers of systemic inflammation specific for HIV-infection (lipopolysaccharide-binding protein; cytokines: IL-1β, IL-6, IL-8, IL-10, TNF -α, INF-γ, INF-α; procalcitonin; inflammatory hsCRP).

All of them will undergo functional testing (Echo, CMR both at rest and stress if necessary) and invasive imaging with QCA, FFR, QFR, OCT, IVUS, VH-IVUS, NIRS.

Patients will be treated according to the current and previous recommendations. Both medical treatment and percutaneous transluminal coronary angioplasty (PTCA) with or without stenting will be done.

Collected data will be analyzed: correlation between ART, blood test results, coronary angiography results, including performed PTCA, history of myocardial infarctions, and other cardiovascular events.

The follow-up period will achieve 12 months prospectively with collected clinical events and imaging outcomes which will be determined at the baseline and 12-month follow-up.

The independent ethics expertise will be provided by the Central Clinical Hospital of the Russian Academy of Sciences (Moscow, Russia). The monitoring of the clinical data with imaging will be provided by The Ethics Board of Central Clinical Hospital of the Russian Academy of Sciences.

DETAILED DESCRIPTION:
HIV, the virus that causes AIDS (acquired immunodeficiency syndrome), is one of the world's most serious health and development challenges. Approximately 38 million people live with HIV, and tens of millions of people have died of AIDS-related causes since the beginning of the epidemic.

However, with increasing access to effective HIV prevention, diagnosis, treatment, and care, including opportunistic infections, HIV infection has transformed from an irreversible terminal illness to chronic disease. Unfortunately, increased life expectancy has increased the risk of other chronic diseases such as cardiovascular diseases (CVD). Actually, CVD has become the most common cause of death in HIV-infected individuals. The risk of myocardial infarction and coronary atherosclerosis prevalence is nearly twice as high in people living with HIV than in the general population. Statins are effective primary prevention for CAD events; however, there are no specific statin use guidelines in HIV. Besides, there is not enough information about systemic inflammation markers and their correlation with atherosclerosis severity.

Nowadays, using invasive imaging, including quantitative coronary angiography with or without further percutaneous coronary intervention, optical coherence tomography/ OCT, intravascular ultrasound/ IVUS, VH-IVUS, near-infrared spectroscopy/ NIRS, cardiovascular events can be predicted and prevented.

In a prospective multicenter observational study, 200 HIV-infected patients treated with antiretroviral treatment (ART) and who suffered from coronary artery disease (CAD) will be enrolled. Blood samples for biological parameters will be collected with all participants: lipid profile and markers of systemic inflammation specific for HIV-infection (lipopolysaccharide-binding protein; cytokines: IL-1β, IL-6, IL-8, IL-10, TNF -α, INF-γ, INF-α; procalcitonin; inflammatory hsCRP).

All of them will undergo functional testing (Echo, CMR both at rest and stress if necessary) and invasive imaging with QCA (Quantitative Coronary Angiography), FFR (Fractional Flow Reserve), QFR (Quantitative Flow Reserve), OCT (Optical Coherence Tomography), IVUS (Intravascular Ultrasound), VH-IVUS (Virtual Histology - IVUS), NIRS (Near Infrared Spectroscopy).

Patients will be treated according to the current and previous recommendations: The 2019 HIV Russian National Guidelines; EACS Guidelines 2020; The AHA scientific statement Characteristics, Prevention, and Management of Cardiovascular Disease in People Living With HIV A Scientific Statement From the American Heart Association. Circulation 2019; ESC/EACTS Guidelines on Myocardial Revascularization 2018; 2019 Guidelines on Chronic Coronary Syndromes.

Both medical treatment and percutaneous transluminal coronary angioplasty (PTCA) with or without stenting will be provided.

The follow-up period will achieve 12 months prospectively with collected clinical events and imaging outcomes which will be determined at the baseline and 12-month follow-up.

The independent ethics expertise will be provided by the Central Clinical Hospital of the Russian Academy of Sciences (Moscow, Russia). The monitoring of the clinical data with imaging will be provided by The Ethics Board of Central Clinical Hospital of the Russian Academy of Sciences.

The clinical data of the HIVE trial include information of the complex examination with:

1. invasive imaging with QCA, FFR, QFR, OCT, IVUS, VH-IVUS, NIRS,
2. two interviews with the risk factor modification recommendations,
3. blood tests:

   * lipid profile (total cholesterol, triglycerides, LDL cholesterol, HDL cholesterol, VLDL cholesterol),
   * markers of systemic inflammation specific for HIV-infection (lipopolysaccharide-binding protein; cytokines: IL-1β, IL-6, IL-8, IL-10, TNF -α, INF-γ, INF-α; procalcitonin; inflammatory hsCRP),
   * biochemical blood test (glucose, asparagine transaminase, alanine transaminase, total bilirubin, creatinine, markers of the myocardium damage (myoglobin, troponin I, creatine kinase, creatine kinase-MB, brain natriuretic peptide - NT-proBNP),
   * complete blood count,
4. ECG,
5. Echo,
6. CMR results

The prospective patients will be tested with HeartAge, SCORE, Duke ACC/ AHA, Duke - DCS, Diamond-Forrester - DFM, The Seattle Angina Questionnaire - SAQ, DukeActivity Status Index -DASI, and EQ-5D-5L, scores that are specific for HIV: EuroSida AIDS/Death risk score, FENCE score, CSRFENCE Score. Patients will be screened for the major risk factors and their modification: unhealthy blood cholesterol levels, high blood pressure, smoking, insulin resistance, diabetes, overweight or obesity, lack of physical activity, unhealthy diet, older age, genetic or lifestyle factors, family history of early heart diseases.

The PCI and PTCA will be undergone by the 2020 ESC/EACTS Guidelines on Myocardial Revascularization. The imaging data from non-invasive (CMR, Echo) and invasive (QCA, FFR, QFR, OCT, IVUS, VH-IVUS, NIRS) methods will be handled and analyzed with the expert-level post-processing imaging software (Medis Suite Solutions: MR, XA, QFR, CT, Intravascular, Ultrasound) from Medis Medical Imaging Systems B.V. (Leiden, The Netherlands).

Our study aims to evaluate the severity of coronary atherosclerosis in HIV-patients with CAD and its correlation with markers of systemic inflammation specific for HIV-infection (LBP; cytokines: IL-1β, IL-6, IL-8, IL-10, TNF -α, INF-γ, INF-α; procalcitonin; inflammatory hsCRP) and to estimate their value in preventing cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* all HIV-positive patients with chronic coronary syndrome or angina equivalent consistent with the manifestation of the stable coronary artery disease (in accordance with the 2019 Guidelines on Chronic Coronary Syndromes);
* patients who underwent CCTA (index procedure) with or without further PCI;
* age above 21 years old;
* patients must receive antiretroviral medications (in accordance to the 2019 HIV Russian National Guidelines; EACS Guidelines 2020);
* lesions may be either de novo or restenotic;
* patient must have one or two-vessel disease in a native coronary vessel requiring or not requiring PCI without indications for immediate bypass surgery with any SYNTAX score;
* successful uncomplicated PCI could be performed in the culprit vessels and all culprit lesions, but there should be no events or complications between the procedures of PCI in the past and 6 months prior to admission to the Chest Pain Center
* the non-culprit vessel should have no flow-limiting lesions (diameter stenosis <39%, but any plaque burden) and must be available for imaging.The non-culprit vessel must be considered safe for imaging evaluation;

Exclusion Criteria:

* any acute comorbidities;
* patient has had a documented ST-elevation acute myocardial infarction within the 24 hours prior to admission to the Chest Pain Center;
* unprotected left main lesion location;
* culprit lesion is located within or distal to an arterial or saphenous vein graft;
* untreated significant coronary lesion with a >50-75% diameter stenosis remaining in the culprit vessel after the planned intervention (branch stenosis is permitted);
* lesion or vessel contains visible thrombus within the imaging procedure;
* patient has an additional lesion that requires intervention within 180 days after the initial hospitalization;
* any diameter stenosis more than 75% in the non-culprit vessel;
* indications for immediate bypass surgery within one year of enrollment with the SYNTAX above 34 (multi-vessel disease requiring intervention in all three major coronary arteries);
* creatinine >150 mmol/L;
* need for dialysis;
* severe endocrine disorders (diabetes is permitted) including pre-existing thyroid diseases;
* decompensated hypotension or heart failure requiring intubation, inotropes,intravenous diuretics, or intra-aortic balloon counterpulsation;
* patient has a known hypersensitivity, allergy, or contraindication to any of the following: aspirin, heparin, clopidogrel, and ticlopidine, or to contrast that cannot be adequately pre-medicated;
* presence of cardiac implants;
* presence of cardiogenic shock;
* patient has a known left ventricular ejection fraction <39%;
* refractory ventricular arrhythmia;
* acute conduction system disease requiring a pacemaker;
* patient has had a recent PCI (last 6 months prior to admission to the Chest Pain Center) unless the patient is undergoing a staged procedure for dual vessel treatment
* prior participation in this study or patient is currently enrolled in another investigational use device, imaging, or drug study that has not been reached its primary endpoint;
* mental diseases, inability for cooperation;
* pregnancy;
* stroke or CVA;
* gastrointestinal bleeding.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All stable chest pain comers with a chronic coronary syndrome without acute angina who underwent QCA, applicable intravascular imaging (OCT, IVUS, VH-IVUS, NIRS) with or without further PCI.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-05 (Actual); Primary Completion 2022-12-05 (Estimated); Study Completion 2023-12-05 (Estimated)

PRIMARY OUTCOMES:
Change of per cent of plaque burden from baseline to follow-up as assessed by QCA | At 12 months after the baseline imaging procedure
  Plaque burden for both culprit and non-culprit lesions will be calculated as a lesion volume (vessel volume-lumen volume)/lumen volume x 1 00. The progression of atherosclerosis and plaque composition in patients receiving different antiretroviral medications will be quantitatively characterized by the parameters of the lesions. The imaging data will be handled with the expert-level post-processing software.
Number of participants with major adverse cardiac events that are related to plaque burden | At 12 months after the baseline imaging procedure
  The composite of cardiac death, cardiac arrest, myocardial infarction, acute coronary syndrome, revascularization by coronary artery bypass surgery (CABG) or percutaneous coronary intervention (PCI), or rehospitalization for angina for patients with both culprit- and non-culprit-lesion-related events. Event rates will be determined at: hospital, at 12months.
Diagnostic value of systemic inflammation markers for risk stratification | At 12 months after the blood testing and the baseline imaging procedure
  To determine prognostic value of systemic inflammation markers (LBP, Lipopolysaccharide binding protein, μg/mL; cytokines: IL-1β, pg/mL; IL-6, pg/mL; IL-8, pg/mL; IL-10, pg/mL; TNF-α, pg/mL; INF-γ, pg/mL; INF-α, pg/mL; procalcitonin, pg/L; inflammatory hsCRP, mg/L) to predict cardiovascular events in patients with HIV.
Invasive assessment of fractional flow reserve for risk stratification | At 12 months after the baseline imaging procedure
  To determine the prognostic value of FFR (fractional flow reserve) when below 0.75-0.80 in comparison with the relevant invasive results of QCA (quantitative coronary angiography), QFR (quantitative flow reserve), OCT (optical coherence tomography), IVUS (intravascular ultrasound), VH-IVUS (virtual histology IVUS), NIRS (near-infrared spectroscopy) handled with the expert-level postprocessing software for predicting cardiac death and nonfatal myocardial infarction.

SECONDARY OUTCOMES:
Change of serologic marker of inflammation CRP from baseline to follow-up | At 12 months after the baseline imaging procedure
  To evaluate a role of HIV and invasive intervention on the inflammatory marker CRP (C-reactive protein, mg/L) as well as its predictive role in comparison with the relevant biochemical variables (LBP, Lipopolysaccharide binding protein, μg/mL; cytokines: IL-1β, pg/mL; IL-6, pg/mL; IL-8, pg/mL; IL-10, pg/mL; TNF-α, pg/mL; INF-γ, pg/mL; INF-α, pg/mL; procalcitonin, pg/L).
Number of participants with procedural success | At 12 months after the baseline imaging procedure
  This is the cumulative variable comprising outcomes of each procedure. Ability to complete the imaging procedures without imaging device or procedure related complication
Change of complexity of coronary artery disease from baseline to follow-up as assessed by SYNTAX score I | At 12 months after the baseline imaging procedure
  Calculated with the version 2.11 of the SYNTAX (Synergy between percutaneous coronary intervention with taxus and cardiac surgery) Score I calculator at: hospital, at 12 months. The variable will be adjusted for CCTA and QCA due to technical limitations. CT SYNTAX score I will be calculated within recommendations Papadopoulou SL, et al, 2013 (JACC Cardiovasc Imaging. 2013 Mar;6(3):413-5. doi: 10.1016/j.jcmg.201 2.09.01 3; http://www.syntaxscore.com/calculator/syntaxscore/frameset.htm; https://syntaxscore2020.com/).
Change of complexity of coronary artery disease from baseline to follow-up as assessed by SYNTAX score II | At 12 months after the baseline imaging procedure
  Calculated with the version 2.11 of the SYNTAX (Synergy between percutaneous coronary intervention with taxus and cardiac surgery) Score II calculator at: hospital, at 12 months. The variable will be adjusted for CCTA and QCA due to technical limitations. CT SYNTAX score II will be calculated within recommendations Papadopoulou SL, et al, 2013 (JACC Cardiovasc Imaging. 2013 Mar;6(3):413-5. doi: 10.1016/ j.jcmg.201 2.09.01 3; http://www.syntaxscore.com/calculator/syntaxscore/framesetss2.htm; https://syntaxscore2020.com/).
Change of fractional flow reserve (FFR) from baseline to follow-up that are related to the progress of atherosclerosis | At 12 months after the baseline imaging procedure
  FFR less than 0.75 considered as hemodynamically significant and estimated for all the lesions. FFR will be compared with other variables to evaluate any correlations.
Change of complexity of coronary artery disease from baseline to follow-up as assessed by Leaman Coronary Score | At 12 months after the baseline imaging procedure
  Calculated within the recommendations of Leaman DM, et al, 1981 (Circulation 63, No. 2, 1981) at: hospital, at 12months. The variable will be adjusted for CTA and 3D QCA due to technical limitations. CT-Leaman score will be calculated within the recommendations of Mushtaq S, et al, 2015 (CircCardiovasc Imaging. 2015 Feb;8(2):e002332.doi: 1 0.11 61 /CIRCIMAGING.11 4.002332).
Number of participants with encephalopathy | At 12 months after the baseline imaging procedure
  The clinical manifestation (medical history, mental status testing with the mini-mental state examination (MMSE) and mini-cog, a physical and neurological exam) of degenerative and/ or paroxysmal encephalopathy will be evaluated with multi-slice computed tomography (MSCT)-screening of the cerebrovascular disease and Alzheimer's disease in association with markers of Herpes Simplex Virus Type 1 (HSV-1 ) and fungi.
Number of chest pain patients with non-obstructive coronary artery disease | At 12 months after the baseline imaging procedure
  Patients with the negative acute markers of the myocardial damage (myoglobin, troponin I, CK, CK-MB, NT-proBNP) and without hemodynamically significant (<50 percent stenosis) coronary atherosclerosis verified by QCA
Number of chest pain patients without coronary artery disease | At 12 months after the baseline imaging procedure
  Patients with the negative acute markers of the myocardial damage (myoglobin, troponin I, CK, CK-MB, NT-proBNP) and without coronary atherosclerosis verified by MSCT

CONTACTS AND LOCATIONS:
Overall Officials: Diana Izimarieva, MD, Principal Investigator — Central Clinical Hospital of the Russian Academy of Sciences; Elena Orlova-Morozova, MD, PhD, Study Director — Moscow Regional Centre For HIV Care and Prevention; Alexey Sozykin, MD, D.Sc, Study Chair — Central Clinical Hospital of the Russian Academy of Sciences; Alexey Nikitin, M.D., D.Sc., Ph.D., Principal Investigator — Central Clinical Hospital of the Russian Academy of Sciences; Eugene Averin, M.D., D.Sc., Ph.D., Principal Investigator — Central Clinical Hospital of the Russian Academy of Sciences; Alexey Shevchenko, M.D., D.Sc., Ph.D., Study Director — Pirogov Russian National Research Medical University
Locations (2):
- Russia (2):
  - Central Clinical Hospital of the Russian Academy of Sciences, Moscow
  - Moscow Regional Centre For HIV Care and Prevention, Moscow

IPD SHARING:
Plan to Share IPD: Undecided
The specific design of the study makes it infeasible to share the required information with the other researchers. Notwithstanding in case of the scientific inquiries regarding meta-analysis the situation might be considered.

REFERENCES:
- See also: Central Clinical Hospital of The Russian Academy of Sciences — https://www.ckbran.ru/en/
- See also: Moscow Regional Centre of HIV Care and Prevention — https://hivmo.ru/